CLINICAL TRIAL: NCT02628418
Title: Feasibility and Efficacy of a Robotic Device for Hand Rehabilitation in Hemiplegic Stroke Patients: a Randomized Pilot Controlled Study
Brief Title: Feasibility and Efficacy of a Robotic Device for Hand Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Palmira Bernocchi, Researcher, Care Continuity Unit, Fondazione Salvatore Maugeri, Institute of Lumezzane, (Brescia), Italy, Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-12-03; First posted 2015-12-11 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Stroke; Upper Extremity Hemiplegia; Disorder of Hand
Keywords: Rehabilitation; Robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gloreha Group (Experimental): The patients in the "Gloreha Group" underwent to following interventions:
  1. General Rehabilitation
  2. Specific hand rehabilitation by Gloreha device
  Interventions: Other: General Rehabilitation; Device: Specific hand rehabilitation by Gloreha device
- Control Group (Other): The patients in the Control Group underwent to following interventions:
  1. General Rehabilitation
  2. Specific hand rehabilitation performed by physiotherapist
  Interventions: Other: General Rehabilitation; Other: Specific hand rehabilitation performed by physiotherapist

INTERVENTIONS:
Other: General Rehabilitation — All patients underwent basic rehabilitation following the guidelines according to the Bobath concept. Mobilization performed by physiotherapist of the lower and upper limbs through passive and/or active manoeuvres, gait training, standing and functional exercises and speech rehabilitation.
Device: Specific hand rehabilitation by Gloreha device — Each training session consisted of six parts:
  1. A sequence of digital joint flexion/extension exercises, from the thumb to the fifth finger (7 min);
  2. 7 min of a number sequence (counting from one to five);
  3. A sequence of thumb-finger opposition movements from the 2nd to the 5th finger (7 min)
  4. A sequence of wave-like finger movements (7 min)
  5. A sequence of fist opening/closing (7 min)
  6. A sequence of flexion-extension of the fingers alternated with flexion-extension of the thumb (5 min).
  Arms: Gloreha Group
Other: Specific hand rehabilitation performed by physiotherapist — The activities were:
  1. Flexion-extension of the fingers (10 min);
  2. Thumb opposition with the other fingers keeping the forearm in supine position (10 min);
  3. Adduction and abduction of the fingers (10 min);
  4. Global movement of the hand consisting in reaching for a 0.5l bottle of water, taking hold of it, pouring water into a glass, and then putting the bottle down and letting go of it (10 min).
  Arms: Control Group

SUMMARY:
Hand recovery following cerebral stroke is complex and requires intensive training. The investigators aimed to evaluate the feasibility and efficacy of robot-assisted hand rehabilitation compared to physiotherapist-guided treatment in recovering dexterity and hand strength in hospitalized sub-acute hemiplegic patients. Design. 30 patients affected by stroke from cerebral ischemia or hemorrhage (Ashworth spasticity index <3) were randomized. Patients in the Treatment group received intensive hand training with Gloreha, a hand rehabilitation glove that provides computer-controlled, repetitive, passive mobilization of the fingers, with multisensory feedback. Patients in the Control group received conventional intensive hand rehabilitation under physiotherapist guidance. Hand motor function (Motricity Index, MI), fine manual dexterity (Nine Hole Peg Test, NHPT) and strength (Grip and Pinch test) were measured at baseline and after rehabilitation, and the differences between final and basal results were compared between groups.

DETAILED DESCRIPTION:
Upper limb recovery, particularly that of the hand, is complex in patients with cerebral stroke and requires an intensive approach.

Regarding upper limb rehabilitation, several research groups have developed robotic devices to provide passive and/or active movements. Their use appears to reduce the motor deficit of the arm and affected hand and to improve hand function both at the wrist and fingers. Hence, the evidence supporting specific robot-assisted rehabilitation of the hand is very promising even if further study is required.In particular, evidence is limited about the benefit of passive exercises and mobilization of the hemiplegic upper limb following stroke, and further research is called for.

In this study the investigators used Gloreha, a new hand rehabilitation glove that provides computer-controlled, repetitive and passive mobilization of the fingers, with multi-sensory feedback. The purpose of the study was to evaluate in the rehabilitation of patients with ischemic or hemorrhagic stroke in the sub-acute phase: 1) the feasibility of this new neuromotor rehabilitation device 2) its efficacy in improving arm function abilities, and 3) the costs involved.

Post-stroke patients admitted for inpatient rehabilitation between May 2013 and January 2014 were screened for enrollment. Eligible patients were randomly assigned, following a simple randomization procedure (computerized random numbers) conducted independently of the study investigators, to Treatment group or Control group, on a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by stroke from cerebral ischemia or hemorrhage that had occurred ≤ 30 days before, with Ashworth spasticity index < 3.

Exclusion Criteria:

* orthopedic limitation (amputations, irreducible articular limitations, advanced osteoarthritis, active rheumatoid arthritis);
* peripheral nerve injury;
* uncontrolled inflammation;
* severe cognitive and behavioral disorders;
* neurodegenerative and neuromuscular diseases;
* Ashworth spasticity index ≥ 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

REFERENCES:
- [Result] Vanoglio F, Bernocchi P, Mule C, Garofali F, Mora C, Taveggia G, Scalvini S, Luisa A. Feasibility and efficacy of a robotic device for hand rehabilitation in hemiplegic stroke patients: a randomized pilot controlled study. Clin Rehabil. 2017 Mar;31(3):351-360. doi: 10.1177/0269215516642606. Epub 2016 Jul 10. PMID 27056250

RESULTS

PARTICIPANT FLOW:
Groups:
- Gloreha Group: The patients in the "Gloreha Group" underwent to following interventions:
  1. General Rehabilitation (GR)
  2. Specific Hand Rehabilitation (SHR) by Gloreha device GR: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept.
  SHR by Gloreha device: Each training session consisted of six parts:
  1.A sequence of digital joint flexion/extension exercises, from the thumb to the fifth finger (7 min); 2.7 min of a number sequence (counting from one to five); 3.A sequence of thumb-finger opposition movements from the 2nd to the 5th finger (7 min) 4.A sequence of wave-like finger movements (7 min) 5.A sequence of fist opening/closing (7 min) 6.A sequence of flexion-extension of the fingers alternated with flexion-extension of the thumb (5 min).
- Control Group: The patients in the Control Group underwent to following interventions:
  1. General Rehabilitation (GR)
  2. Specific hand rehabilitation performed by physiotherapist (SHR) GR: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept.
  SHR performed by physiotherapist: The activities were:
  1. Flexion-extension of the fingers (10 min);
  2. Thumb opposition with the other fingers keeping the forearm in supine position (10 min);
  3. Adduction and abduction of the fingers (10 min);
  4. Global movement of the hand consisting in reaching for a 0.5l bottle of water, taking hold of it, pouring water into a glass, and then putting the bottle down and letting go of it (10 min).
Period: Overall Study
Arm/Group | Gloreha Group | Control Group
Started | 15 | 15
Completed | 14 | 13
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Gloreha Group: The patients in the "Gloreha Group" underwent to following interventions:
  1. General Rehabilitation (GR)
  2. Specific Hand Rehabilitation (SHR) by Gloreha device
  GR: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept. Mobilization performed by physiotherapist of the lower and upper limbs through passive and/or active manoeuvres, gait training, standing and functional exercises and speech rehabilitation.
  SHR by Gloreha device: Each training session consisted of six parts:
  1. A sequence of digital joint flexion/extension exercises, from the thumb to the fifth finger (7 min);
  2. 7 min of a number sequence (counting from one to five);
  3. A sequence of thumb-finger opposition movements from the 2nd to the 5th finger (7 min)
  4. A sequence of wave-like finger movements (7 min)
  5. A sequence of fist opening/closing (7 min)
  6. A sequence of flexion-extension of the fingers alternated with flexion-extension of the thumb (5 min).
- Control Group: The patients in the Control Group underwent to following interventions:
  1. General Rehabilitation
  2. Specific Hand Rehabilitation (SHR) performed by physiotherapist
  General Rehabilitation: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept. Mobilization performed by physiotherapist of the lower and upper limbs through passive and/or active manoeuvres, gait training, standing and functional exercises and speech rehabilitation.
  SHR performed by physiotherapist: The activities were:
  1. Flexion-extension of the fingers (10 min);
  2. Thumb opposition with the other fingers keeping the forearm in supine position (10 min);
  3. Adduction and abduction of the fingers (10 min);
  4. Global movement of the hand consisting in reaching for a 0.5l bottle of water, taking hold of it, pouring water into a glass, and then putting the bottle down and letting go of it (10 min).
- Total: Total of all reporting groups
Arm/Group | Gloreha Group | Control Group | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (11) | 73 (14) | 72.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Completed the Hand Rehabilitation Program
Time Frame: Through study completion. The specific hand interventionn consisted of a total of 30 sessions, lasting 40 min/day, for 5 days/week , from admission to discharge in the Rehabilitation Centre, over a period of about 6 weeks.
Measure: Number; unit: participants
Arm/Group | Gloreha Group | Control Group
Number analyzed (Participants) | 15 | 15
participants | 14 | 13

2. Primary Outcome: Side Effects Using Gloreha Device
Description: The feasibility of the device was assessed in terms of side effects (the physiotherapist was required to report any adverse events occurring during the study in regard to the use of Gloreha);
Time Frame: Through study completion. The specific hand intervention consisted of a total of 30 sessions, lasting 40 min/day, for 5 days/week , from admission to discharge in the Rehabilitation Centre, over a period of about 6 weeks.
Measure: Number; unit: side effects
Groups:
- Gloreha Group: The patients in the "Gloreha Group" underwent to following interventions:
  1. General Rehabilitation (GR)
  2. Specific Hand Rehabilitation (SHR) by Gloreha device GR: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept.
  SHR by Gloreha device: Each training session consisted of six parts:
  1. A sequence of digital joint flexion/extension exercises, from the thumb to the fifth finger (7 min);
  2. 7 min of a number sequence (counting from one to five);
  3. A sequence of thumb-finger opposition movements from the 2nd to the 5th finger (7 min)
  4. A sequence of wave-like finger movements (7 min)
  5. A sequence of fist opening/closing (7 min)
  6. A sequence of flexion-extension of the fingers alternated with flexion-extension of the thumb (5 min).
Arm/Group | Gloreha Group | Control Group
Number analyzed (Participants) | 14 | 13
side effects | 0 | 0

3. Primary Outcome: Efficacy in Improving Arm Function Abilities Measured by the Change From Baseline in Motricity Index at End of Inpatient Rehabilitation
Description: Motricity Index, a measure of the motor function of the paretic upper limb. Motricity Index used to measure the ability to activate a muscle group to move a body segment through a range of motion and resist external force. The upper extremity motricity index includes: 1. pinch grasp, 2. elbow flexion, and 3. shoulder abduction.
  The total upper extremity score involved adding one to the sum of the three actions.
  The score of each action ranges from 0 (no ability) to 33 (maximal ability) with a maximum possible score=100.
Time Frame: Baseline and end of the study after 30 sessions, an average of 6 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Control Group: The patients in the Control Group underwent to following interventions:
  1. General Rehabilitation
  2. Specific hand rehabilitation performed by physiotherapist
  General Rehabilitation: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept. Mobilization performed by physiotherapist of the lower and upper limbs through passive and/or active manoeuvres, gait training, standing and functional exercises and speech rehabilitation.
  Specific hand rehabilitation performed by physiotherapist: The activities were:
  1. Flexion-extension of the fingers (10 min);
  2. Thumb opposition with the other fingers keeping the forearm in supine position (10 min);
  3. Adduction and abduction of the fingers (10 min);
  4. Global movement of the hand consisting in reaching for a 0.5l bottle of water, taking hold of it, pouring water into a glass, and then putting the bottle down and letting go of it (10 min).
Arm/Group | Gloreha Group | Control Group
Number analyzed (Participants) | 14 | 13
units on a scale | 23.0 [13.6 to 32.4] | 5.2 [-0.4 to 10.7]

4. Primary Outcome: Efficacy in Improving Arm Function Abilities Measured by the Change From Baseline in Nine Hole Peg Test at End of Inpatient Rehabilitation.
Description: Nine Hole Peg Test (NHPT), a measure of coordination and mono-manual dexterity. It consists in collecting 9 pegs and inserting them into holes in a wooden base within a 50-sec time limit. The score is the average number of pegs inserted/tests performed.
Time Frame: Baseline and end of the study after 30 sessions, an average of 6 weeks
Measure: Mean (95% Confidence Interval); unit: pegs/sec
Groups:
- Control Group: The patients in the Control Group underwent to following interventions:
  1. General Rehabilitation (GR)
  2. Specific hand rehabilitation (SHR) performed by physiotherapist GR: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept.
  SHR on performed by physiotherapist: The activities were:
  1. Flexion-extension of the fingers (10 min);
  2. Thumb opposition with the other fingers keeping the forearm in supine position (10 min);
  3. Adduction and abduction of the fingers (10 min);
  4. Global movement of the hand consisting in reaching for a 0.5l bottle of water, taking hold of it, pouring water into a glass, and then putting the bottle down and letting go of it (10 min).
Arm/Group | Gloreha Group | Control Group
Number analyzed (Participants) | 14 | 13
pegs/sec | 0.16 [0.09 to 0.25] | 0.02 [-0.02 to 0.07]

5. Secondary Outcome: The Feasibility of This New Neuromotor Rehabilitation Device (Gloreha)
Description: The feasibility of the device was assessed in terms of the level of operator difficulty for the physiotherapist in managing the device, assessed by visual analogue scale (VAS) (0 extremely simple - 10 extremely difficult). This outcome was measured only in the Gloreha Group in which patients were treated with device.
Time Frame: Baseline and end of the study after 30 sessions, an average of 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gloreha Group
Number analyzed (Participants) | 14
units on a scale | 3.15 (1.0)

6. Secondary Outcome: Efficacy in Improving Arm Function Abilities Measured by the Change From Baseline in Grip Test at End of Inpatient Rehabilitation.
Description: The Grip test is a measure of hand strength. Each patient, at baseline and at the end of the study, repeated the test 3 times and the mean value was normalized for body mass index (BMI).
Time Frame: Baseline and end of the study after 30 sessions, an average of 6 weeks
Measure: Mean (95% Confidence Interval); unit: kg / (kg / m ^ 2)
Groups:
- Control Group: The patients in the Control Group underwent to following interventions:
  1. General Rehabilitation (GR)
  2. Specific hand rehabilitation (SHR) performed by physiotherapist GR: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept.
  SHR performed by physiotherapist: The activities were:
  1. Flexion-extension of the fingers (10 min);
  2. Thumb opposition with the other fingers keeping the forearm in supine position (10 min);
  3. Adduction and abduction of the fingers (10 min);
  4. Global movement of the hand consisting in reaching for a 0.5l bottle of water, taking hold of it, pouring water into a glass, and then putting the bottle down and letting go of it (10 min).
Arm/Group | Gloreha Group | Control Group
Number analyzed (Participants) | 14 | 13
kg / (kg / m ^ 2) | 0.27 [0.13 to 0.41] | 0.03 [-0.005 to 0.07]

7. Secondary Outcome: Efficacy in Improving Arm Function Abilities Measured by the Change From Baseline in Pinch Test at End of Inpatient Rehabilitation.
Description: The Pinch test is a measure of hand strength. Each patient, at baseline and at the end of the study, repeated the test 3 times and the mean value was normalized for body mass index (BMI).
Time Frame: Baseline and end of the study after 30 sessions, an average of 6 weeks
Measure: Mean (95% Confidence Interval); unit: kg / (kg / m ^ 2
Groups:
- Gloreha Group: TThe patients in the "Gloreha Group" underwent to following interventions:
  1. General Rehabilitation (GR)
  2. Specific Hand Rehabilitation (SHR) by Gloreha device GR: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept.
  SHR by Gloreha device: Each training session consisted of six parts:
  1.A sequence of digital joint flexion/extension exercises, from the thumb to the fifth finger (7 min); 2.7 min of a number sequence (counting from one to five); 3.A sequence of thumb-finger opposition movements from the 2nd to the 5th finger (7 min) 4.A sequence of wave-like finger movements (7 min) 5.A sequence of fist opening/closing (7 min) 6.A sequence of flexion-extension of the fingers alternated with flexion-extension of the thumb (5 min).
- Control Group: The patients in the Control Group underwent to following interventions:
  1. General Rehabilitation (GR)
  2. Specific hand rehabilitation (SHR) performed by physiotherapist. GR: All patients underwent basic rehabilitation following the guidelines according to the Bobath concept.
  SHR performed by physiotherapist: The activities were:
  1. Flexion-extension of the fingers (10 min);
  2. Thumb opposition with the other fingers keeping the forearm in supine position (10 min);
  3. Adduction and abduction of the fingers (10 min);
  4. Global movement of the hand consisting in reaching for a 0.5l bottle of water, taking hold of it, pouring water into a glass, and then putting the bottle down and letting go of it (10 min).
Arm/Group | Gloreha Group | Control Group
Number analyzed (Participants) | 14 | 13
kg / (kg / m ^ 2 | 0.07 [0.03 to 0.1] | 0.02 [-0.001 to 0.04]

8. Secondary Outcome: Efficacy in Improving Arm Function Abilities Measured by the Change From Baseline in Quick-DASH Questionnaire at End of Inpatient Rehabilitation.
Description: The Arm disability was assessed of the study with the Quick version of the Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) questionnaire.
  The Quick-DASH is a 19-item ordinal scale with a 5-level rating of items from 1 (no difficulty) to 5 (unable to do).
  Quick-Dash can be divided into an 11-item (abilities and symptoms) and an 8-item optional work module and sports/performing arts module. In the 11-item sub-scale, the subject defines the ability to perform some actions (8 items) and the intensity of some symptoms (3 items), referring to the previous week. The total score range is from 19 (no disability) to 95 (full disability).
Time Frame: Baseline and end of the study after 30 sessions, an average of 6 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gloreha Group | Control Group
Number analyzed (Participants) | 14 | 13
units on a scale | -15.7 [-25.7 to 5.8] | -0.43 [-4.5 to 3.6]

9. Secondary Outcome: The Costs Involved in Using Gloreha in the Rehabilitation
Description: Costs were calculated in terms of the time required by healthcare personnel, using the average cost per hour of a physiotherapist per total number of rehabilitation treatments per patient. The equivalent cost of the device for the period of patient treatment was calculated incorporating depreciation, considering the estimated residual value of the device with depreciation rate of 20%.. Indirect costs were not considered because these were common to both groups.
Time Frame: Through study completion, from admission to discharge in the Rehabilitation Centre, over a period of about 6 weeks.
Measure: Number; unit: Euros/patient
Arm/Group | Gloreha Group | Control Group
Number analyzed (Participants) | 14 | 13
Euros/patient | 237 | 480

ADVERSE EVENTS:
Time Frame: Through study completion, from admission to discharge in the Rehabilitation Centers, over a period of about 6 weeks.
Description: Three patients lost to follow-up for clinical problems not for side effects related to SHR. If Gloreha was able to open a spastic hand it would be potentially dangerous (the glove was not sensitized) so we cannot know exactly what happens on the patients' hand. If the force applied by Gloreha was such as to open a spastic hand it could cause pain.
Arm/Group | Gloreha Group | Control Group
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gloreha Group (N=15) | Control Group (N=15)
Bacterial infection (Infections and infestations) | 0 (0) | 2 (2)
Rheumaoid arthitis (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No